CLINICAL TRIAL: NCT02678910
Title: Ovarian Tissue Freezing For Fertility Preservation In Women Facing A Fertility Threatening Medical Diagnosis Or Treatment Regimen
Brief Title: Ovarian Tissue Freezing For Fertility Preservation In Women Facing A Fertility Threatening Medical Diagnosis/Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vlad Radulescu (Other)
Responsible Party: Sponsor-Investigator, Vlad Radulescu, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-0927-F1V
Record Dates: First submitted 2014-05-08; First posted 2016-02-10 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Cancer; Hematologic Disorder; Rheumatologic Disorder; Infertility
MeSH Terms: conditions — Neoplasms; Hematologic Diseases; Collagen Diseases; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ovarian Cryopreservation (Experimental): Removal of the ovary for cryopreservation is an investigational procedure. 100% of the tissue will be used for the participant's future use.
  Interventions: Procedure: Ovarian Cryopreservation

INTERVENTIONS:
Procedure: Ovarian Cryopreservation — The ovarian tissue will be removed at a UK Healthcare facility and evaluated for gross disease by a pathologist, embryologist, andrologist or REI physician. The ovarian cortex will be dissected from the medulla and cut into strips in culture/holding media, washed to remove blood cells, and cryopreserved. Cryopreservation will be performed using modifications of the techniques described by Gosden et al. (1994) or will be vitrified using a modification of the techniques of Kuwayama et al., 2007.

SUMMARY:
The purpose of this research is to obtain ovarian tissue from female participants who will receive therapy which is expected to result in a loss or impairment of ovarian function and/or infertility and wish to preserve (freeze) ovarian tissue for the purpose of initiating a pregnancy in the future.

Removal of the ovary for cryopreservation is an investigational procedure. 100% of the tissue will be used for the participant's future use. There have been 86 pregnancies as a result of frozen ovarian tissue that has been re-implanted back into the pelvis and hormonal function has been restored in individuals for up to 7 years.

By doing this study, the investigators hope to learn of how to successfully freeze and thaw ovarian tissue in a manner that permits subsequent use by patients at some point in the future. Participation may also advance our knowledge of how to successfully mature follicles and oocytes (eggs) that are contained in these tissues which may help others in the future.

DETAILED DESCRIPTION:
The research procedures will be conducted at the University of Kentucky (UK) Medical Center.

Participants in the study will provide ovarian tissue cryopreservation for their own personal use.

The duration of the study will be until the participant reaches age 41 years. Participants will be broken out into four categories:

Participants will have surgical removal of their ovarian tissue using the methods determined by their surgeon based on their medical/surgical diagnosis or treatment. Participants in one of the following categories will participant in the study:

1. Participants have elected to have one or both ovaries removed for the treatment or prevention of disease.
2. Participants who have elected to have surgery to remove all or part of one or both ovaries for medical reasons where cryopreservation of the remaining limited portions of normal ovarian cortex is the only option for fertility preservation at the time (except that ovarian cortex from the ovary that contains the mass will not be cryopreserved).
3. Participants who have elected to have surgery to remove all or part of one or both ovaries for medical reasons where cryopreservation of the remaining limited portions of normal ovarian cortex is the only option for fertility preservation at the time but who cannot or will not provide tissue to the research pool (except that ovarian cortex for the ovary that contains the mass will not be cryopreserved).
4. Participants who have elected to have one or part of one ovary removed, solely for the purpose of fertility preservation because they are not candidates for or choose not to use more mature fertility preservation technologies.

Participants undergoing elective removal of an ovary (category C above) will undergo a procedure called laparoscopy to remove the ovary. This surgery will be performed under general anesthesia and one ovary will be removed in total through an instrument channel employing standard techniques of operative laparoscopy. This surgical procedure is performed solely for fertility preservation but will potentially be coordinated with another procedure such as placement of a central line for future chemotherapy or laparotomy for another purpose. Although only one ovary will be removed, both of the participant's ovaries must appear normal for the procedure to be completed. The ovary to be removed will be chosen at the time of surgery based on appearance and ease of removal. After the surgery is complete, the participant will not have any further procedures except for a routine post-operative visit. A 0.5 cm cross section from the short axis of the ovary will be provided to the Department of Pathology for routine histological evaluation, and the remaining tissue will be processed for cryopreservation. If pathology finds evidence of cancer in the ovarian tissue provided at surgery, they may request that all of the participant's tissue (even tissue that has been frozen for their use) be returned to pathology for a more detailed examination. In this case, no tissue is available for the participant to use for fertility preservation purposes.

b. Cryopreservation: Ovarian tissue will be cryopreserved under the protocol originally established by the National Physicians Cooperative of the Oncofertility Consortium. The ovarian tissue will be removed at a UK or Norton Healthcare facility and evaluated for gross disease by a pathologist, embryologist, andrologist or a reproductive endocrinology and infertility (REI) physician. The ovarian cortex will be dissected from the medulla and cut into strips in culture/holding media, washed to remove blood cells, and cryopreserved. Cryopreservation will be performed using modifications of the techniques described by Gosden et al. (1994) or will be vitrified using a modification of the techniques of Kuwayama et al., 2007. The procedure for cryopreservation/vitrification may be modified as improvements become available.

The designated laboratory directors at UK responsible for the overall quality of the ovarian tissue cryopreservation.

c. Tissue storage: Cryopreserved participant tissues will be transferred to Reprotech, Ltd (RTL) in Roseville, Minnesota for storage and subsequent release. Reprotech, Ltd. is an FDA compliant and American Association of Tissue Banks accredited long term storage facility for reproductive tissues. Based on the extended periods of time that these tissues are likely to be stored Reprotech, Ltd. provides maximum flexibility for the participants involved. In this way, the participant can store tissues as long as they wish and ship them to a fertility treatment center of their choice at the time of use. The participant can determine how her own tissue will be used as technology changes and based on her unique circumstances. Reprotech, Ltd. does not perform fertility treatments and is not affiliated with any fertility center so there is no potential conflict of interest.

d. Infectious Disease Screening and Testing: Banking and subsequent use of ovarian tissue is regulated by the Food and Drug Administration (FDA). In order to comply with current tissue banking regulations and to be prepared for any future changes in regulations while these ovarian tissues are in storage, participants will be tested and screened for a number of infectious diseases prior to banking ovarian tissue.The testing will include but not be limited to testing for Hepatitis B and C and HIV. The testing that will be performed will be testing that is mandated for donors of leukocyte rich tissues and must be performed within 7 days of tissue procurement. In this way, the tissue could potentially be used by the participant herself and it could also be suitable for use in another individual (such as a surrogate) in the future if indicated by the participant's medical diagnosis.

If the ovarian tissue was vaginally removed during surgery the sites will also collect a vaginal swab from the participant for Gonorrhea and Chlamydia testing.

Please note that if the HIV screening test is positive, a confirmatory test will then be performed. Should the screening tests detect that participants are infected with HIV this information will be communicated confidentially to them through personal contact by a qualified professional. Participants will meet with a qualified professional who will provide HIV counseling.

There are risks associated with this study and those risks are outlined in the study informed consent document.

Benefit vs. Risk: There is no guarantee that participants will get any benefit from taking part in this study, although 86 babies have been born from transplanted frozen ovarian tissue. A females participation may provide her with a means to restore her fertility and reproductive hormonal function in the future as observed in previous reports. A females participation may also advance the investigator's understanding of how to successfully freeze and thaw ovarian tissue in a manner that permits subsequent use by the participant and other patients at some point in the future. A females participation may also advance the investigator's knowledge of how to successfully mature follicles and oocytes (eggs) that are contained in these tissues which may help the participant or others in the future. However, there is a significant possibility that there may be no direct benefit to the participant from her participation in this research study. Specifically, there is the possibility that ovarian cryopreservation will not result in successful pregnancy in the future.

There are alternatives to taking part in this study and those alternatives are addressed in the study informed consent document.

Costs: All expenses related to the research procedure will be covered by the research funds and include the oophorectomy, anesthesia, pathologist's fees and infectious disease testing.

Either the participant or their insurance company, Medicare or Medicaid will be responsible for the costs of all care and treatment that the participant would receive during this study that she would normally receive for her condition. These are costs that are considered medically reasonable and necessary and will be part of the care she receives if she does not take part in this study. This includes the confirmatory HIV testing and the follicle stimulating hormone (FSH) testing.

There are also costs associated with the handling, processing, shipping and storage of ovarian tissue. Those costs are outlined in the study informed consent document.

In the unlikely event that the participant is hurt or injured while participating in this study the medical costs related to their care and treatment will be their responsibility or submitted to their insurance.

ELIGIBILITY:
Inclusion Criteria:

* Undergo standard of care surgery, chemotherapy, drug treatment, and/or radiation for the treatment or prevention of a medical condition or malignancy expected to result in permanent and complete loss of subsequent ovarian function.
* Or, have a medical condition or malignancy that requires removal of all or part of one or both ovaries.
* May have newly diagnosed or recurrent disease. Those who were not enrolled at the time of initial diagnosis are eligible if they have not received therapy that is viewed as likely to result in complete and permanent loss of ovarian function.
* Participant undergoing elective removal of an ovary for fertility preservation only must have two ovaries.
* Participant who already has stored cryopreserved ovarian tissue in a frozen state prior to undergoing cancer treatments (surgery, chemotherapy or radiation) will be eligible for enrollment with informed consent.
* Is not a candidate for or chooses not to utilize embryo or oocyte banking.

Exclusion Criteria:

* Psychological, psychiatric or other conditions which prevent giving fully informed consent.
* Underlying medical condition which significantly increases risk of complications from anesthesia and surgery.
* Participants with a large cancerous mass in the ovary that is being removed; cryopreservation will not be performed on portions of the ovary.
* Blood testing indicates that the participant does not have enough eggs remaining in her ovary.

Ages: 12 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Number of subjects who elect to have ovarian tissue cryopreservation in one year. | 1 year from IRB protocol approval and study open date
  The investigator will describe the number of subjects who elect ovarian tissue cryopreservation (OTC) over a 1 year period of time to determine feasibility of OTC in oncology subjects receiving chemotherapy and radiation.

SECONDARY OUTCOMES:
Number of subjects who elect to have ovarian tissue cryopreservation over a 5 year prior period of time. | 5 years from IRB protocol approval and study open date
  The investigator will describe the number of subjects who elect ovarian tissue cryopreservation (OTC) over a 5 year period of time to determine feasibility of OTC in oncology subjects receiving chemotherapy and radiation.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Wagner, MD, Study Director — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - Norton Health Care, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: No